CLINICAL TRIAL: NCT00466362
Title: One Year Observational Study on Effects of Lifestyle Intervention in Morbidly Obese Persons With Type 2 Diabetes.
Brief Title: Lifestyle Intervention in Obesity, Effect on Diabetes
Status: Withdrawn | Type: Observational
Why Stopped: Recruitment problems
Sponsor: Tor-Ivar Karlsen (Other)
Responsible Party: Sponsor-Investigator, Tor-Ivar Karlsen, RN, Evjeklinikken
Organization: Evjeklinikken (Other)
Other Study IDs: EK0702
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Type 2 Diabetes
Keywords: Obesity; Diabetes; Weight; Lifestyle; Follow up
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Diabetes Mellitus; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: The Evje Model — Lifestyle intervention

SUMMARY:
There are evidence from numerous studies on effect of lifestyle intervention in morbidly obese patients with type 2 diabetes. This study examines the effect of the "Evje-model" on type 2 diabetes.

The "Evje-model" is a combined 12 months model, consisting of repeated stays in a specialist centre, telephone follow-up at home, home groups, self monitoring and close contact with the patients' local physician.

DETAILED DESCRIPTION:
There will be done QOL-measures, blood- and urine analysis, weight, waist- and hip measurement, blood pressure and VO2-max measurement at baseline, after 6 months and after 12 months.

ELIGIBILITY:
Inclusion Criteria:

* All patients with BMI > 35 with diagnosed type 2 diabetes
* Referred to Lifestyle Intervention from a public hospital

Exclusion Criteria:

* Pregnancy
* Active major psychiatric disease(s)
* Active and serious eating disorder
* Drug- and/or alcohol dependency

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Morbidly obese patients
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-04; Primary Completion 2008-01 (Actual); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life | 2007

CONTACTS AND LOCATIONS:
Overall Officials: Tom B Schulz, Dr. Med., Principal Investigator — Evjeklinikken
Locations (1):
- Evjeklinikken AS, Evje Og Hornnes, Evjemoen, Norway